CLINICAL TRIAL: NCT04740372
Title: Development of an International Questionnaire to Assess Patient-reported Quality of Life Related to COVID-19 Disease, the Oslo COVID-19 Quality of Life Questionnaire (QLQ) - ## © Phase III of Questionnaire Development
Brief Title: Development of an International COVID-19 Specific Quality of Life Questionnaire, Phase III. The OSLO COVID-19 QLQ
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Medical University Innsbruck (Other); Johannes Gutenberg University Mainz (Other); Servicio de Navarro de Salud (Unknown); University of Southampton (Other); Skane University Hospital (Other); Haukeland University Hospital (Other); University of the East Ramon Magsaysay Memorial Medical Center (Unknown); Sumandeep Vidyapeeth (Other); Birzeit University (Unknown); National Centre for Infectious Diseases (Unknown); Komfo Anokye Teaching Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Delphin Amdal, Head of PROMiNET, Research support service, Oslo University Hospital
Other Study IDs: REK Norway: 171640
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Covid19, Patient Reported Outcome Measures, Quality of Life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. Method study. Psychometric testing — Patients will fill in the questionnaire followed by an interview (phase IIIA) or a debriefing questionnaire (Phase IIIB)

SUMMARY:
Purpose: to develop an international validated patient-reported outcome measure for COVID-19 patients according to international guidelines.

In this phase III of the project, the preliminary questionnaire of 80 items will be tested. It has been developed based on literature review and interviews with health care professionals and patients (phase I-II).

In Phase III A patients will fill in the questionnaire followed by interviews on relevance, importance and wording of the questionnaire In Phase III B patients will fill in the questionnaire and an debriefing questionnaire. We will do explorative psychometric analyses.

DETAILED DESCRIPTION:
This project aim to develop an international validated patient-reported outcome measure for COVID-19 patients according to international guidelines. The Phase I and II of this development process have been finalized. Based on a systematic literature review , interviews with 44 health-care professionals and 52 patients in 6-7 countries a final list of 80 questions, the preliminary Oslo COVID-19 QLQ - PW80 ©, is ready to be tested in the current Phase III of the development process.

The objectives of the phase III are:

* In a limited patient group, to check that the items make sense to the target population, that the phrasing and sequence of questions is acceptable, that there are no missing issues and that none of the questions are confusing and/or offensive (Phase IIIA).
* In addition, in a larger patient group, to test hypothesized subscales for psychometric properties including reliability, prevalence and variance (e.g. Cronbach's alpha coefficient and correlation-based methods) (Phase IIIB).

The end-product, the international COVID-19- specific questionnaire, will be a psychometrically robust patient-reported outcome measure (PROM) to assess HRQoL in patients with or after COVID-19 disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with verified SARS-CoV-2 infection (positive test according to local/national standards)
* Patients with active or previous symptomatic COVID-19 disease
* In-patients in hospitals and nursing homes or out-patients in hospitals or patients discharged from institutions to their home/covid-19 centres or patients staying at home/covid-19 centres during the course of the disease
* Patients aged 18 years and older
* Ability to read and comprehend the process and study documents as judged by the investigator
* Written informed consent

Exclusion Criteria:

* Patients in intensive care units (can be recruited after they have been dismissed)
* Inability to read and comprehend the process and study documents as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To ensure content validity of the final questionnaire, the participants will be recruited according to specified recruitment matrices based on countries, language groups, age, gender, hospitalisation status, disease status and comorbidity.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Validated COVID-19 specific questionnaire | 6 months
  Instrument that can be used in international intervention and observational studies on patients with COVID-19 disease

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amdal CD, Falk RS, Singer S, Pe M, Piccinin C, Bottomley A, Appiah LT, Arraras JI, Bayer O, Buanes EA, Darlington AS, Arbanas GD, Hofso K, Holzner B, Sahlstrand-Johnson P, Kulis D, Parmar G, Rmeileh NMEA, Schranz M, Sodergren S, Bjordal K. A multicenter international prospective study of the validity and reliability of a COVID-19-specific health-related quality of life questionnaire. Qual Life Res. 2023 Feb;32(2):447-459. doi: 10.1007/s11136-022-03272-2. Epub 2022 Oct 23. PMID 36273365
- See also: The questionnaire is available at Mapi Research Trust — https://eprovide.mapi-trust.org/advanced-search?search=COVID-19%20QLQ